CLINICAL TRIAL: NCT01498627
Title: Cervarix Long-term Safety Surveillance Using the PGRx Information System (PGRx Study)
Brief Title: Cervarix Long-term Safety Surveillance
Acronym: PGRx
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112677
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: Infections, Papillomavirus
Keywords: Autoimmune diseases (AIDs); Cervarix; PGRx information system
MeSH Terms: conditions — Papillomavirus Infections; Autoimmune Diseases | interventions — human papillomavirus vaccine, L1 type 16, 18; Data Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Case Group: Subjects in this group are incident cases (i.e. newly diagnosed subjects) reported as having occurred in the previous twelve months before the recruitment consultation.
  Interventions: Biological: Cervarix; Other: Data collection
- Control Group: Subjects selected from the pool of potential referents reported by physicians in general practice, who meet the same general inclusion and exclusion criteria as the cases.
  Interventions: Biological: Cervarix; Other: Data collection

INTERVENTIONS:
Biological: Cervarix — 3 doses over a period of 6 months (Month 0 and ideally Month 1 and Month 6, with 1 month minimum between any two doses).
Other: Data collection — PGRx information system

SUMMARY:
This study aims to assess whether the use of Cervarix® is associated with a modified risk of central demyelination, type 1 diabetes (DT1), Cutaneous Lupus, inflammatory arthritis, idiopathic thrombocytopenic purpura (ITP), Lupus erythematosus, myositis and dermatomyositis, Guillain-Barre syndrome and/or Autoimmune thyroiditis and Graves disease by using the PGRx information system.

DETAILED DESCRIPTION:
PGRx is an information system that intends to bridge the resource gap to assess the effect of a drug on the risk of adverse events that are infrequent and/or with a long delay of onset. It uses some characteristics of the ad hoc case-control or case-referent design, transposed on a prospective, on-going, population-based recruitment plan. This particular design is called here systematic case-referent design in contrast to the ad hoc case-control or case-referent methodology. The PGRx information system is based on the routine and targeted recruitment of cases of a series of pathologies, compared to population-based referents for the study of exposure to a wide variety of drugs. Drug exposure ascertainment is obtained from two different sources in the PGRx.

system: A) A structured patient interview (telephone-administered questionnaire) B) The medical data form with the computerized medical prescriptions (interview guide)

ELIGIBILITY:
Inclusion Criteria:

* Male and female
* Age 14 to 79 years-old (included)
* Patient residing in France
* Patient accepting to participate in the study
* Patient can read and respond to a telephone interview

Exclusion Criteria:

* Prior reported history of the disease
* Patient or Patient's parent cannot read the interview guide or answer a telephone interview questionnaire in French
* Refusal to participate

Ages: 14 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects reporting an Autoimmune diseases (AID) in the previous 12 months before recruitment consultation and those whose AID is reported by physicians in general practice
Sampling Method: Non-Probability Sample
Enrollment: 2945 (Actual)
Dates: Start 2008-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To assess whether the use of Cervarix® is associated with a modified risk of central demyelination. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of type 1 diabetes. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of cutaneous Lupus. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of inflammatory arthritis. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of idiopathic thrombocytopenic purpura. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of systemic lupus erythematosus. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of addendum for cutaneous lupus. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of myositis. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of dermatomyositis. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of Guillain-Barrre syndrome. | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of autoimmune thyroiditis | At Month 36
To assess whether the use of Cervarix® is associated with a modified risk of Graves disease. | At Month 36

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline